CLINICAL TRIAL: NCT06686628
Title: An Open-label, Drug-drug Interaction Study to Investigate the Effects of Amlitelimab on the Pharmacokinetics of Selected Cytochrome P450 Substrates in Adult Participants With Moderate-to-severe Atopic Dermatitis
Brief Title: An Open-label, DDI Study to Investigate the Effects of Amlitelimab on the PK of Selected Cytochrome P450 Substrates
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT18404; U1111-1303-3406 (Registry Identifier: ICTRP); 2024-513495-17 (Registry Identifier: CTIS)
Record Dates: First submitted 2024-11-11; First posted 2024-11-13 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Dermatitis Atopic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Midazolam; Caffeine; Metoprolol; Omeprazole; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Amlitelimab and CYP substrates (Experimental): A single oral dose of a CYP450 substrates cocktail which will include caffeine, metoprolol, midazolam, omeprazole, and warfarin will be administered.
  A single dose of amlitelimab will then be administered on several days. A single oral dose of CYP450 substrates cocktail in combination with the last single dose of amlitelimab.
  Interventions: Drug: Amlitelimab; Drug: Midazolam; Drug: Caffeine; Drug: Metoprolol; Drug: Omeprazole; Drug: Warfarin

INTERVENTIONS:
Drug: Amlitelimab — Pharmaceutical form: Injection solution Route of administration: SC injection
  Other Names: SAR445229
Drug: Midazolam — Pharmaceutical form: Solution Route of administration: Oral
Drug: Caffeine — Pharmaceutical form: Tablet Route of administration: Oral
Drug: Metoprolol — Pharmaceutical form: Tablet Route of administration: Oral
Drug: Omeprazole — Pharmaceutical form: Capsule Route of administration: Oral
Drug: Warfarin — Pharmaceutical form: Tablet Route of administration: Oral

SUMMARY:
This is an open-label, single group, 2-period, Phase 1, single-sequence study. The study duration will be up to 342 days. The treatment period will be up to Week 29, where Week 29 is defined as End of Treatment (last amlitelimab administration at Week 25).

The number of visits will be 23 or 21 visits for participants who decide to continue amlitelimab therapy in the long-term extension study LTS17367 (RIVER-AD) study.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

* Male or female participant aged 18 to 65 years (inclusive), at the time of the informed consent is signed.
* Participants must have AD as defined by the American Academy of Dermatology Consensus Criteria (2014) for 1 year or longer before signing of informed consent.
* The EASI score ≥16 at Screening and Check-in (Day -1).
* vIGA-AD score ≥3 (on the 0 to 4 vIGA-AD scale) at Screening and Check-in (Day -1).
* AD involvement of ≥10% body surface area at Screening and Check-in (Day -1).
* Participants must have documented history within 6 months prior to Screening and Check-in (Day -1), of either inadequate response (including inadequate efficacy or medical inadvisability) of topical treatments.
* Body weight within 40 to 150 kg at Screening and Day 1 and body mass index (BMI) <40 kg/m2 (inclusive).
* Capable of giving signed informed consent.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Known history of significant immunosuppression or suspected current significant immunosuppression, including history of invasive opportunistic, or helminthic infections.
* Any malignancies or history of malignancies prior to baseline (except for non-melanoma skin cancer that has been excised and cured for more than 5 years prior to baseline).
* Any concomitant illness that would, in the Investigator's opinion, inhibit the participant's participation in the study, including for example, but not limited to, hypertension, renal disease, neurological conditions, heart failure, and pulmonary disease.
* Any medical condition which, in the Investigator's opinion may present an unreasonable risk to the study participants as a result of his/her participation in this clinical study, may make participant's participation unreliable, or may interfere with study assessments.
* Any active or chronic infection including helminthic infection requiring systemic treatment within 4 weeks prior to baseline (1 week in the event of superficial skin infections) and any infection which as per Investigator's opinion precludes the participant's participation in the study or acute infection requiring treatment with systemic antibiotics, antivirals, antiprotozoals, or antifungals at Screening or Check--in (Day -1).
* History or presence of substance abuse (including alcohol, nicotine) prior to Check-in (Day 1/V2) or regular alcohol consumption (>14 units per week for males and >7 units per week for females).
* In the Investigator's opinion, medical conditions related to prior AD medications that have not healed/fully recovered for more than 2 weeks before the Screening visit, including, but not limited to, conjunctivitis, keratitis, eosinophilic conditions, arthralgia, herpes zoster, thrombosis.
* Use of tobacco- or nicotine-containing products within 6 months prior to Check-in (Day -1).
* Poor metabolizers for CYP2C9, CYP2C19, or CYP2D6 based on genotyping.
* Treatment with a live (attenuated) vaccine within 12 weeks prior to baseline; failure to complete non-live immunization required by local regulation (eg, vaccination for COVID-19) at least 14 days prior to baseline.
* Any contraindication to one or more of the following CYP cocktail study interventions, according to the applicable labeling:

  * Caffeine
  * Metoprolol
  * Midazolam
  * Omeprazole
  * Warfarin
* Administration, within 14 days before baseline or within a period of 5 times the elimination half-life of the medication before baseline, whichever is longer, of any medication that is a known inducer or inhibitor of either one or more of the following CYP enzymes: CYP3A4, CYP2C19, CYP2C9, CYP2D6, and CYP1A2.
* Administration, within 14 days before baseline or within a period of 5 times the elimination half-life of the medication before baseline, whichever is longer, of:

  * Caffeine
  * Metoprolol
  * Midazolam
  * Omeprazole
  * Warfarin.
* Consumption of any 1 or more of the following food items and/or beverages within 1 week prior to baseline:

  * Grapefruit or grapefruit juice, apple or apple juice, orange or orange juice, lemons or lemon juice, limes or lime juice
  * Vegetables from the mustard green family (eg, broccoli)
  * Charbroiled meats
  * Caffeinated beverages, foods or drugs containing caffeine as well as decaffeinated coffee.

Participants who are not willing to abstain from the consumption of these food items and/or beverages for certain periods during the study (Day 1 to Day 8, and Day 168 to Day 183) will also be excluded.

* History of excessive consumption of beverages containing caffeine (more than 4 cups or glasses per day). Participants who are not willing to abstain from the consumption of caffeine within 1 week prior to baseline, Day 1 to Day 8, and Day 168 to Day 183 will also be excluded.
* Female participants who are using any form of hormonal contraceptives (eg, oral, injectables, implants, patches, rings, hormone-impregnated IUDs) for birth control.
* Have previously completed or withdrawn from this study or any other study investigating amlitelimab or have previously received a dose of an investigational drug within the past 90 days or 5 half-lives, whichever is longer, prior to Check-in (Day -1).
* Concurrent participation in any other clinical study, including non-interventional studies.
* Participants positive for human immunodeficiency virus; participants with any of the following results at Screening (Visit 1): presence of HBsAg with or without HBV DNA PCR test or presence of antibody to hepatitis B core antigen (HBcAb) or presence of antibody to HBsAg with positive HBV DNA PCR test; positive hepatitis C total antibody confirmed by positive Hepatitis C virus RNA.
* Known or suspected hypersensitivity to any of the study interventions (amlitelimab, CYP substrates [cocktail compounds]) or excipients, or drug or other allergy that, in the opinion of the Investigator, contraindicates participation in the study.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-11-21 (Actual); Study Completion 2026-04-03 (Estimated)

PRIMARY OUTCOMES:
AUC and AUClast for CYP substrates | Baseline (Day 1 to Day 8) and Day 176 to Day 183
  AUC = area under the serum/plasma concentration curve; AUClast = area under the plasma concentration versus time curve calculated using the trapezoidal method from time zero to the real time tlast.

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events, serious adverse events, adverse event of special interest, and potentially clinically significant abnormality. | Baseline through Day 316
Serum amlitelimab concentrations (Ctrough) measured. | Day 8 through Day 316
  Ctrough = plasma concentration pre-dose
Tmax, t1/2z, and tlast of CYP substrates alone and co-administered with amlitelimab | Baseline (Day 1 to Day 8) and Day 176 to Day 183
  tmax = time to reach the maximum plasma concentration observed t1/2z = terminal half-life associated with the terminal slope tlast= time corresponding to the last concentration above the limit of quantification
Cmax of CYP substrates alone and co-administered with amlitelimab | Baseline (Day 1 to Day 8) and Day 176 to Day 183
  Cmax = maximum plasma concentration observed.
Incidence of anti-drug antibodies of amlitelimab. | Baseline through Day 316

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational Site Number : 2760001, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: INT18404 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26214&tenant=MT_SNY_9011